CLINICAL TRIAL: NCT03095898
Title: Electroacupuncture Analgesia for Colonoscopy: A Prospective and Randomized Study
Brief Title: Electroacupuncture Analgesia for Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Fady Daniel, Assistant Professor, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IM.FD.05
Record Dates: First submitted 2017-03-02; First posted 2017-03-30 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Colonoscopy; Acupuncture
Keywords: Colonoscopy; Acupuncture
MeSH Terms: interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- True Acupuncture (Experimental)
  Interventions: Device: Electroacupuncture
- Sham Acupuncture (Sham Comparator)
  Interventions: Device: Electroacupuncture
- Control Group (No Intervention)

INTERVENTIONS:
Device: Electroacupuncture — Acupuncture is a form of alternative medicine and is used worldwide for different indications, mainly for pain management. It relies on the stimulation of specific acupuncture points along the skin of the body using thin needles.
  Arms: Sham Acupuncture; True Acupuncture

SUMMARY:
The objective of this study is to compare the effectiveness of acupuncture versus Sham acupuncture in reducing patient's discomfort and pain during colonoscopy with a standard sedation protocol. This will be objectively measured by the reduction in the amount of analgesia used as well as the time spent in the recovery room.

DETAILED DESCRIPTION:
Aim of the study

The objective of this study is to compare the effectiveness of acupuncture versus Sham acupuncture in reducing patient's discomfort and pain during colonoscopy with a standard sedation protocol. This will be objectively measured by the reduction in the amount of analgesia used as well as the time spent in the recovery room.

Background and significance

Colonoscopy is an invasive procedure, known to be uncomfortable for patients, necessitating the use of sedative drugs. The standard practice at the institution is to use conscious sedation with midazolam and fentanyl to achieve a satisfactory level of relaxation, cooperation, and amnesia during the procedure. Patients undergoing colonoscopy might experience abdominal cramps, pain and distension necessitating an increase in the sedation used in most of the times, in addition to aborting the procedure in rare cases. Previous studies have reported that the use of sedative and analgesic drugs frequently prolongs recovery room observation and brings rare but well-known adverse events like hypotension and respiratory compromise. To note that the former complications of conscious sedation are dependent on the doses of drugs used.

Acupuncture is a form of alternative medicine and is used worldwide for different indications, mainly for pain management. It relies on the stimulation of specific acupuncture points along the skin of the body using thin needles. It is based on the belief that a "life force" circulates within the body in lines called meridians. Each meridian corresponds to an internal organ. Only few publications exist with respect to the role of acupuncture for sedation during gastrointestinal procedures. These studies showed that that the stimulation of LI4, S36, SP6 and SP9 acupuncture points can decrease the demand for sedative drug, as well as gastrointestinal discomfort and pain by electrically stimulating bilateral active points.Sham acupuncture on the other hand uses analogous stimulation of inactive symmetrical points near the active points.

A similar study found a decrease in both frequency and intensity of post-procedural abdominal pain, abdominal distension , along with a shorter duration in the recovery room, however, the study didn't assess the decrease in the sedation requirements between the different groups.

Another study showed that the time to pass the sigmoid and splenic flexure and time to reach the cecum were significantly shorter in the acupuncture group compared to the control group.

The researchers hypothesize that "true" acupuncture or sham acupuncture can have an analgesic and a sedative effect that will lead to a reduction of the dosage of midazolam or fentanyl needed for satisfactory sedation during colonoscopies.

Research design and methods:

This study is designed as a single center, randomized, sham controlled trial. To test this hypothesis the researchers will compare three groups. Group 1 will receive true-acupuncture at the traditional acupuncture points P6, SP9, ST36, LI4; group 2 will get sham-acupuncture and group 3 will be the control group without any acupuncture needle insertion. All three groups will receive standard sedation with midazolam/fentanyl as it is the standard practice at the institution. To note, that the sedation requirements are dependent on patients and physician preferences. The endoscopist performing the procedure will be blinded to the randomization.

The acupuncture will be performed by a qualified staff physician, and the patients enrolled in group A will have acupuncture bilaterally on the upper arms and lower legs as per the following points:

1. LI4 (Hegu, the 4th point on the Large Intestine channel), on the dorsum of the hand, between the first and second metacarpal bones, at the midpoint of the second metacarpal bone, and close to its radial border.
2. S36 (Zusanli, the 36th point on the Stomach channel), below the knee, one-finger breadth lateral to the anterior crest of the tibia, three-finger breadth inferior to the hollow that is formed below the patella, and lateral to the patellar ligament when the knee is flexed.
3. SP9 (Yinlingquan, the 9th point on the Spleen channel), on the medial side of the lower leg, in a depression in the angle formed by the medial condyle of the tibia and the posterior border of the tibia.
4. P6 (Nei Guan, the 6th point on pericardium channel) is located three finger breadths below the wrist on the inner forearm in between the two tendons.

I. Patient Recruitment

This study will take place at the endoscopy unit of the American University of Beirut Medical center. Eligible patients for participation in this clinical trial are those planned to undergo elective diagnostic or therapeutic colonoscopy under midazolam/fentanyl sedation, aged above 18 years, and ASA (American Society of Anaesthesiology) classification I-III, who give written informed consent. After checking the inclusion and exclusion criteria, the participant will be approached in the clinic by the primary physician or someone responsible for his clinical care to inform him about the study. After gaining the participant's permission to participate in the study, the participant will be approached by Mrs. Ghada Shami, the Registered Nurse responsible for explaining the preparation for colonoscopy will screen for interested patients. She will then notify the divisional research fellow, Dr Mahmoud Rahal to further explain the study concept and details to these patients in a private setting in the clinics area.

II- Primary endpoints:

Primary endpoint of the study is the used dosage of midazolam, in combination with fentanyl.

III- Secondary endpoints:

Secondary endpoint is patients' and gastroenterologists' satisfaction with the procedure, determined with a visual analog scale, from 0 to 10. The researchers will also compare the time needed to complete the procedure and the time spent in the recovery room, between all three groups.

V- Study Plan

After the patient has signed the informed consent form, randomization will be performed as a permuted block randomization. Allocation to treatment group will be performed by sealed consecutively numbered envelopes. One experienced and qualified staff acupuncturist (Dr Fadila Nagi) will perform the intervention in the preparation room. Needles inserted will be disposable and single use. The participants will be connected to a portable electro-stimulator and left in place for 20 min. The intervention with electroacupuncture will be stopped after 20 mins and the colonoscopy will start afterwards.

In group A, the true acupuncture group, the needles will be placed in the following points, which are considered relevant both - for sedation and for abdominal distension: Pericardium 6 (P6), Spleen 9 (SP9) ,Stomach 36 (ST36), and Large intestine 4 (LI4).

In group B, patients will receive Sham-acupuncture with the same sort of needles. The needles will be placed 2-3 cm distal and lateral to the used acupoints (P6, ST36, and LI4) on locations that are not known as acupuncture points. The electrostimulator to be used in the study is "AS SUPER 4 digital" made in Germany with a frequency of 2 Hz, pulse width 210 microseconds alternating with 15 Hz, pulse width 120 microseconds. Aiming to reach an intensity of 3 mA.

In group C, the control group, patients will not have any needles inserted.

Patients will be monitored using SpO2, heart rate and noninvasive blood pressure measurements as it is usually performed prior, during and after each colonoscopy.

The risks associated with this study are minimal. The needles used will be single use, this is why there is no associated infectious risk; however, participants might experience minimal pain and small hematomas at the acupuncture needle insertion site and some patients might experience vasovagal reaction from the needle insertion. The risks concerning the electrical stimulation of acupuncture needles are limited to mildly uncomfortable muscle twitching around the sites of needle insertion at the level of the hands and legs. If acupuncture proves to be able to reduce the required amounts of sedative drugs employed during colonoscopy, this will translate into a better patient tolerance of the procedure and potentially less associated cardio-vascular and pulmonary side effects.

VI-Sample size calculation and data analysis:

The sample size calculation was in fact done after determining the median doses of Midazolam and fentanyl administered in the endoscopy unit during a 3 months period. Dr Hani Tami was the statistician consulted. The average fentanyl dose is 73, and the standard deviation is 24. Accordingly, to detect a 20% reduction (which is 15 units), and a standard deviation of 24, 42 patients are needed in each group (total is multiplied by 3), to detect this difference, at an 80% power and 0.05 error. As for the midazolam, average is 4.3 and standard deviation is 1.6, and accordingly, 55 patients in each group is needed to detect a 20% reduction, and a total of 165 patients will be needed. The sample size was then increased to 180 for each group to allow for possible dropouts.

VII-Funding for the Study

Dr. Fady Daniel will generously provide the acupuncture needles needed for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects undergoing colonoscopy as part of their clinical care
2. midazolam/fentanyl sedation
3. age above 18 years
4. ASA classification I-III,
5. Able to give written informed consent

Exclusion Criteria:

1. Age < 18 years
2. ASA classification VI and V
3. Allergic reaction to planned medication in the patients' medical history
4. Nickel allergy
5. Pacemaker/Implanted Cardioverter Device
6. Psychiatric and neurologic disorders including epilepsy
7. Use of anticoagulants and antiplatelet including aspirin
8. Previous colonic resection,
9. Patients refusing conscious sedation
10. Active GI bleeding
11. Patients who had any technical knowledge of acupuncture were also excluded to maintain blindness between acupuncture and sham acupuncture
12. Patients with arrhythmia
13. Patients with skin disorders in the vicinity of electrodes placement
14. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-01-09 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-02-15 (Estimated)

PRIMARY OUTCOMES:
Reduction in amount of analgesia | 1 day per patient
  Used dosage of midazolam, in combination with fentanyl

SECONDARY OUTCOMES:
Patients and gastroenterologist satisfaction | 1 day per patient
  Patients and gastroenterologist satisfaction using Visual Analog Scale (0-10)
Time needed to complete the procedure | 1 day per patient
  Time needed to complete the procedure using Minutes:Seconds
Time spent in the recovery room | 1 day per patient
  Time spent in the recovery room using Minutes:Seconds

CONTACTS AND LOCATIONS:
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No